CLINICAL TRIAL: NCT00311350
Title: Ascending Multiple Dose Study of the Safety, Tolerability, and Pharmacokinetics of MOA-728 Administered Orally to Healthy Subjects
Brief Title: Study Evaluating the Safety of MOA-728 Administered Orally to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Jeff Cohn, Salix Pharmaceuticals
Allocation: Randomized | Masking: Double
Other Study IDs: 3200A3-100
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Postoperative Complications; Constipation
Keywords: Safety; Health; Pharmacokinetics; ileus
MeSH Terms: conditions — Postoperative Complications; Constipation; Ileus

INTERVENTIONS:
Drug: MOA-728

SUMMARY:
This is the first multiple-dose experience in humans with MOA-728 in an oral formulation. This study will provide an assessment of the safety, tolerability, and pharmacokinetics (PK) of MOA-728 following administration of ascending multiple oral doses to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48
Dates: Start 2006-03; Study Completion 2006-08

PRIMARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Cohn, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Philadelphia, Pennsylvania, United States